CLINICAL TRIAL: NCT06141759
Title: The Effect of Schroth Best Practice Exercises and Cheneau Brace Treatment on Perceptual and Cognitive Asymmetry in Adolescent Idiopathic Scoliosis With Thoracic Major Curve
Brief Title: The Effect of Conservative Treatment on Perceptual and Cognitive Asymmetry in Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, Assistant professor, Bandırma Onyedi Eylül University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bandırma University
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Schroth Best Practice Exercises and Cheneau braces. There were 18 sessions, each lasting 90 minutes, a total of 6 weeks for the exercise training.
  Interventions: Other: Exercise
- Control Group (No Intervention): For six weeks, no application was made.

INTERVENTIONS:
Other: Exercise — Cheneau brace and Schroth Best Practice exercise
  Arms: Intervention group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) patients have been found to exhibit cortical asymmetry. This study aimed to examine the impact of conservative treatments on perceptual and cognitive asymmetry in the auditory system assessed by dichotic listening in AIS patients with thoracic major curves.

DETAILED DESCRIPTION:
Background: Adolescent idiopathic scoliosis (AIS) patients have been found to exhibit cortical asymmetry. This study aimed to examine the impact of conservative treatments on perceptual and cognitive asymmetry in the auditory system assessed by dichotic listening in AIS patients with thoracic major curves. Method: This study involved 30 AIS patients and 21 healthy subjects. The intervention group used a Cheneau brace and performed 18 Schroth Best Practice (SBP) exercise sessions. Auditory lateralization was assessed using the Dichotic Listening Paradigm (DLP) in both groups before and after the intervention.

ELIGIBILITY:
Inclusion Criteria for Intervention Group:

* Having been diagnosed with AIS,
* Being 10-16 years of age,
* Having a Cobb angle of between 20° and 50°
* Risser's sign of 0-3,
* Having right thoracic scoliosis,
* Being right-handed,
* Having received no previous treatment that may affect scoliosis,
* Having no chronic disease requiring the use of medication.

Inclusion Criteria for Intervention Group:

* Participants aged 10-16 years

Exclusion Criteria for both groups:

* Having previous spinal operations,
* Hearing loss, or the presence of other muscular, neurological, or rheumatic diseases.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Dichotic Listening Paradigm | 6 weeks
  The Dichotic Listening Paradigm is a method that provides behavioral information to determine auditory system asymmetry and is reliable for use with adolescents. The DLP was implemented in both groups at baseline and at the end of week 6 in a seated position with eyes open in a quiet room. In this paradigm, syllables ba, da, ga, pa, ta, and ka were utilized; these were standardized by the Dokuz Eylül University Music Sciences Voice Studio for Turkish society

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Burçin Akçay, Balıkesir
  - Bandırma Onyedi Eylül University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Balıkesir

REFERENCES:
- [Derived] Akcay B, Inanc G. The effect of Schroth Best Practice exercises and Cheneau brace treatment on perceptual and cognitive asymmetry in adolescent idiopathic scoliosis with thoracic major curve. Ir J Med Sci. 2024 Jun;193(3):1479-1486. doi: 10.1007/s11845-023-03593-2. Epub 2023 Dec 20. PMID 38123885